CLINICAL TRIAL: NCT03618199
Title: Efficacy of a Transcranial Vibrating System for Minimizing Dizziness During Caloric Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Olith10101
Record Dates: First submitted 2018-07-24; First posted 2018-08-07 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Vestibular Function Tests; Dizziness
Keywords: Caloric testing; vestibular nystagmography; VNG; Videonystagmography
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: First phase: test 20 subjects. They will undergo the "caloric testing" part of the standard vestibular testing, with and without our transcranial vibration system (10 with device on then off, 10 with device off then on) and will describe their state on a "visual analog scale" (both dizziness and nausea) at the end.
  Success is 1) substantially reduced dizziness ad nausea, 2) statistically unchanged clinical measures.
  If (and only if) the first phase is successful, we proceed to the second phase.
  Second phase: identical to first phase, but is conducted with patients coming in the clinic for vestibular testing. The order ("device on" first, or second) will be randomly assigned.
Who Masked: Outcomes Assessor
Masking Description: Subject in both phases will immediately know whether the transcranial vibrating system is on. Analysis of outcomes (1-dizziness, 2-nausea, 3-clinical measures from vestibular nystagmography resulting from the caloric testing) will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Efficacy of vibrating system on healthy volunteers (Experimental)
  Interventions: Device: Efficacy of transcranial vibrating system on mitigating dizziness and nausea during caloric testing
- Efficacy of vibrating system on vestibular patients (Experimental)
  Interventions: Device: Efficacy of transcranial vibrating system on mitigating dizziness and nausea during caloric testing

INTERVENTIONS:
Device: Efficacy of transcranial vibrating system on mitigating dizziness and nausea during caloric testing — Transcranial vibrating system will be on then off (or off then on in a random order) during a repeated application of the "calorics testing" stimulus, i.e. warm or cold water irrigated in the left (then right) ear canal. The effect of the vibrating system on 1) resulting dizziness and nausea often experienced by patients and 2) clinical parameters measured by caloric testing will be quantified.

SUMMARY:
Vestibular disorders are among the most common causes of disability in society. Vestibular dysfunction affects over one third of the population over the age of 40 and a significant percentage of the younger population. Vestibular disorders have a dramatic impact on daily life impacting work, relationships, and even activities of daily living. Diagnosis of vestibular disorders is often facilitated by functional vestibular tests. The most common of these tests is videonystagmography, during a critical portion of which, the "caloric test," warm and cool stimuli are presented in the outer ears to stimulate the inner ear vestibular system. The vertigo produced by caloric stimulation not uncommonly results in nausea, and sometimes vomiting, sometimes to the point of not being able to complete the test protocol. In this project we examine a device that has shown promise and might be beneficial for improving the testing for vestibular disorders. We hypothesize that with this device, the nausea associated with caloric testing will be significantly reduced when the device is used, while it will not change the results of the test in a statistically significantly manner.

To date, the device has only been systematically tested on healthy volunteers.

DETAILED DESCRIPTION:
Vestibular disorders can be difficult to diagnose and can vary in symptoms and fluctuate in severity. It is typically hard to determine which vestibular system (left/right) might be causing the vestibular disorder, as both sides normally work in unison. Testing the vestibular function in each side (left/right) of a patient is typically done with "caloric testing", which allows testing the left and right vestibular systems separately. However, it leads to nausea in most patients, and part of the clinical test is spent waiting for the patient to recover. Many patients undergoing caloric testing experience nausea to the point that some patients cannot complete the test, while others need a long period of time to recover from the nausea and dizziness induced by the testing. While it is hoped that this project will ultimately help establish the effectiveness of the transcranial vibration system for a range of vestibular disorders, we choose caloric testing for an initial assessment because it is performed daily in the clinic, it is easy to administer, and there is very little controversy about its use.

Specific Aims: Using Otolith Labs' device, we wish:

1. To determine if subjects undergoing caloric testing treated with the device

   1. Experience less nausea than with no device, or
   2. If the subjects do experience nausea, whether the time to resolution is shorter with the device than with no device.
2. To determine if the clinical results obtained by caloric testing are significantly different with the device compared to not wearing the device.

Objectives:

Primary: To demonstrate the efficacy of a bone conduction device at preventing nausea in subjects undergoing vestibular (particularly caloric) testing, as measured by the reduction from baseline of symptoms associated with (caloric)-testing

Secondary: To show that the use of the bone conduction device does not change the clinical measures obtained by vestibular caloric testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject can speak and comprehend English.
2. Subject can stand a strap placed on their head for an hour.

Exclusion Criteria:

1. History of head injury within the last six months
2. Presence of severe aphasia
3. History of diagnosed neuropsychiatric disorders
4. Documented neurodegenerative disorders
5. Pregnancy [Female candidates will be asked if they are pregnant]
6. History of Cerebrovascular disorders
7. History of ear operation other than myringotomy and tube placement in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Nausea and dizziness | VAS administered ten minutes post-caloric testing; data will be analyzed upon study completion, estimated to last 6 weeks
  Visual Analog Scales (VAS, adapted from "Visual Vertigo Analogue Scale" for dizziness and "Baxter Retching Faces (BARF)" for nausea) will be filled out by the subject ten minutes after each phase of the caloric testing, i.e. "with" and "without" the transcranial vibration system. Each phase of the caloric testing itself takes approximately 30 minutes. These Visual Analog Scales range from 0 to 10 (None to Agonizing). They will provide independent measures of the effectiveness of the transcranial vibration system.

SECONDARY OUTCOMES:
Vestibular testing outcomes | Vestibular clinical measures will be analyzed by a clinician upon study completion, estimated to last 6 weeks.
  Nystagmus associated with caloric testing (the primary clinical measure derived from caloric testing) will be compared, in the "with device" and "without device" conditions.

CONTACTS AND LOCATIONS:
Overall Officials: David J Eisenman, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No